CLINICAL TRIAL: NCT03411733
Title: Prevalence of Helicobacter Pylori in Patients With Acne Vulgaris
Brief Title: Prevalence of H.Pylori in Patients With Acne Vulgaris Acne Vulgaris
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Dina Ali, Resident physician, Department of Dermatology, Sohag Educational Hospital, Sohag University
Other Study IDs: HPAV001
Record Dates: First submitted 2018-01-20; First posted 2018-01-26 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Helicobacter Pylori Infection; Acne Vulgaris
Keywords: acne vlugaris; prevalence; Helicobacter Pylori
MeSH Terms: conditions — Acne Vulgaris | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and stool samples were retained for a short period (few hours) till completion of laboratory analyses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acne vlugaris group: Included recruited patients with acne vulgaris Intervention: Blood and stool samples collection
  Interventions: Other: Blood and stool samples collection
- Control group: Included healthy participants Intervention: Blood and stool samples collection
  Interventions: Other: Blood and stool samples collection

INTERVENTIONS:
Other: Blood and stool samples collection — Collection of blood and stool samples from each participants for H.pylori antigen/ antibody detection

SUMMARY:
The objective of the study is to investigate prevalence of H.Pylori infection among acne vulgaris patients.

DETAILED DESCRIPTION:
The study included patients with acne vulgaris and healthy control participants. The study recruited both sexes, all grades of acne, adolescents and young adults.

All patients were subjected to complete history, general and skin examination Acne vlugaris Patients were classified into mild, moderate and severe according to the classification of American Academy of dermatology for acne vulgaris.

Detection of H. pylori infection:

Blood and stool samples were taken from each participant and was directly transferred to laboratory for detection of H. Pylori antigen and antibody.

An enzyme-linked immune sorbent assay (ELISA) was used for quantitative assessment of IgG antibodies against H.Pylori in human serum.

A monoclonal antibodies based enzyme-linked immunosorbent assay was used to detect H.Pylori specific antigen in stool samples.

ELIGIBILITY:
Inclusion Criteria:

* Acne vulgaris patients
* Healthy volunteers (control)

Exclusion Criteria:

* Patients with a history of drug intake that affects H. Pylori such as proton-pump inhibitors, clarithromycin, tetracyclines, amoxicillin or metronidazole within previous two weeks were excluded.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with acne vulgaris and presented to Dermatology outpatient clinic, Sohag University hospital.
  Healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
H.pylori infection | one year
  Prevalence of H.pylori infection among acne group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan Saleh, MD, Study Director — Sohag Faculty of Medicine
Locations (1):
- Dermatology outpatient clinic, Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
All available data shall be shared with other researchers upon their request after agreement of study director